CLINICAL TRIAL: NCT02510859
Title: Nutrition and Life QUality Patients With Head and Neck Cancers
Acronym: NUQUE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-101
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systematic nutritional consultation at home (Experimental): Patients will be followed by a dietician at the patient's home at weeks 2 (S2) and 4 (S4) of radiotherapy, then at the end of radiotherapy at T0. Monitoring will be continued 15 days after the end of irradiation and then one month (T1 and 2 months (T2). A personalized follow will be performed and a document entitled "Dietary own program" will be given to the patient.
  Interventions: Other: Systematic nutritional consultation at home
- Traditional nutritional follow up (No Intervention): Traditional nutritional follow up that is to say with a nutritional consultation before starting treatment and then when necessary on medical advice

INTERVENTIONS:
Other: Systematic nutritional consultation at home — Patients will be followed by a dietician at the patient's home at weeks 2 (S2) and 4 (S4) of radiotherapy, then at the end of radiotherapy at T0. Monitoring will be continued 15 days after the end of irradiation and then one month (T1 and 2 months (T2). A personalized follow will be performed and a document entitled "Dietary own program" will be given to the patient.
  Arms: Systematic nutritional consultation at home

SUMMARY:
Malnutrition is currently a major factor of morbidity and mortality, which poses a major public health problem in developing countries but also, albeit to a lesser degree and for different reasons, for industrialized countries. It is recognized that in countries "of the North", from 30 to 60% of hospitalized patients suffer from dénutrition.

In any case, it is covered by an imbalance between the contributions and needs; the two main mechanisms are a delivery failure (fasting, ingesting difficulty ...) and / or increased requirements (hypermetabolism ...). In cancer patients the Aero-Digestive Upper Airways (VADS), this imbalance is even more pronounced than the two mechanisms exist and potentiate. Patients included in this study are a population at risk, because of their therapeutic containing at least radiotherapy. It is recognized that this form of therapy exposes dental complications, mucous, saliva. These complications have a deleterious effect on the nutritional status of patients.

The diagnosis, treatment and prevention of dénutritions have an important place in the therapeutic strategies of this type of cancer because it is events whose incidence and morbid consequences are high and for which there are appropriate nutritional treatments in most cas. While the complete correction of malnutrition generally passes by the effective etiological treatment of the causal pathology, therapeutic efficacy of the latter is often conditioned by the nutritionnel state.

In addition to these concepts, investigators wants to study the benefits of a diet followed during the irradiation phase of patients with head and neck cancers and New treaties. We propose a randomized, phase III, open, multicenter, to evaluate the impact of a dietary consultation at home on the life quality of patients with head and neck cancer including first therapeutic sequence involves radiotherapy more or less aware. The duration of the study is 24 months.

The main objective is to evaluate the impact of a dietary consultation at home on the life quality of patients with head and neck cancer including first therapeutic sequence involves a more or less sensitized radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years
* having Given written consent
* Life span > 3 months
* Score WHO <3
* Patient With cancer of Aero-Digestive tract Superior histologically proven (including salivary glands)
* Stable , presenting no other progressive neoplasia except VADS
* Patient to be treated with radiotherapy alone or concomitant chemoradiotherapy or radiotherapy with cetuximab or postoperative radiotherapy roughly sensitized.
* Patient Fluent French.

Exclusion Criteria:

* Patient with history of malignancy, except basal cell cancer or neck cancer treated and cured
* Patient who underwent salvage surgery other than a course node,
* Patient with other evolutionary neoplasia at the time of examination
* Patient having previously had a mutilating surgery (causing effects on swallowing and feeding)
* Uncontrolled infectious disease
* Lactating or pregnant women or lack of contraception in reproductive years
* Intercurrent pathology involving life-threatening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2010-12; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
EVA score "Quality of Life = overall mental and social physical condition at the time of the interview" | after 3 months of the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Service ORL et de chirurgie cervico- faciale, Caen CHU, France